CLINICAL TRIAL: NCT02984657
Title: Evaluation of Operating Room Reverse Trendelenburg Positioning and Its Effect on Postoperative Hypoxemia, Aspiration, and Length of Stay: a Retrospective Study of Consecutive Patients
Brief Title: Reverse Trendelenburg Positioning and Its Effect on Outcomes: a Retrospective Study of Consecutive Patients
Status: Completed | Type: Observational
Sponsor: C. Michael Dunham (Other)
Collaborators: St. Elizabeth Youngstown Hospital (Unknown)
Responsible Party: Sponsor-Investigator, C. Michael Dunham, Research Associate, St. Elizabeth Youngstown Hospital, Mercy Health Ohio
Organization: Mercy Health Ohio (Other)
Other Study IDs: 15-023
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Aspiration, Respiratory; Hypoxia; Perioperative Period; Supine Position
Keywords: Hypoxemia; Reverse Trendelenburg
MeSH Terms: conditions — Respiratory Aspiration; Hypoxia; Deception | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2012 patients: Surgical patients in 2012 with anesthesia and nursing staff less attuned to intraoperative RTP.
  Interventions: Procedure: Surgical patients in 2012 with anesthesia and nursing staff less attuned to intraoperative RTP.
- 2015 patients: Surgical patients in 2015 with enhanced anesthesia and nursing staff awareness and use of intraoperative RTP.
  Interventions: Procedure: Surgical patients in 2015 with enhanced anesthesia and nursing staff awareness and use of intraoperative RTP.

INTERVENTIONS:
Procedure: Surgical patients in 2012 with anesthesia and nursing staff less attuned to intraoperative RTP. — RTP, reverse Trendelenburg positioning
  Groups: 2012 patients
Procedure: Surgical patients in 2015 with enhanced anesthesia and nursing staff awareness and use of intraoperative RTP. — RTP, reverse Trendelenburg positioning
  Groups: 2015 patients

SUMMARY:
The purpose of this study is to investigate whether intraoperative reverse Trendelenburg positioning decreases postoperative hypoxemia and perioperative pulmonary aspiration rates.

DETAILED DESCRIPTION:
Intraoperative pulmonary aspiration can cause death and lead to morbidity. In addition, reliable estimates of aspiration rates are uncertain. In part, this ambiguity relates to the lack of prospective data. Relevant studies are retrospective chart reviews or results from voluntary reporting databases. Furthermore, aspiration diagnosis can be imprecise. The finding is certain when there is aspiration of bile or particulate matter from the tracheobronchial tree or there is endoscopic visualization. However, the diagnosis is presumptive when there is intraoperative or postoperative development of a new chest x-ray infiltrate and attendant tachypnea, hypoxia, wheezing, or changes in ventilator airway pressures.

Most patients undergoing general endotracheal anesthesia are in the supine or horizontal position. However, evidence from the literature demonstrates that the supine position in mechanically ventilated patients is a risk for aspiration and ventilator associated pneumonia (VAP). During intensive care unit (ICU) mechanical ventilation, the Institute for Healthcare Improvement recommends elevating the head of the bed to prevent pulmonary aspiration and VAP. Other investigations have shown a profound relationship between horizontal positioning and intra-operative aspiration. There is substantial operating room, ICU, and animal investigative evidence that aspiration occurs despite the presence of a cuffed endotracheal tube. Likewise, previous work by this group showed a 30% perioperative hypoxemia rate, which was significantly associated with horizontal positioning. The post-operative length of hospital stay was 2 days longer with hypoxemia, compared to no hypoxemia (p <0.0001) and this represented a total of 300 additional days for the 2 months of the study.

The purpose of this retrospective study is to repeat the investigation after adopting a recent policy change of 10-degree Reverse Trendelenburg position as the routine for surgical patients, unless deemed inappropriate by either the anesthesiology or operating room nursing staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endotracheal intubation and general anesthesia
* Age ≥18 years
* Glasgow Coma Scale score ≥13 (prior to tracheal intubation)
* American Society of Anesthesiologists classification I-IV
* Pre-operative pulmonary stability

Exclusion Criteria:

* Tracheal intubation prior to emergency department arrival
* Cardiac and thoracic surgical patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients from an urban hospital
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postoperative hypoxemia | 48 hours postoperatively

SECONDARY OUTCOMES:
Perioperative pulmonary aspiration | 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Dunham, MD, Principal Investigator — St. Elizabeth Youngstown Hospital
Locations (1):
- St. Elizabeth Youngstown Hospital, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunham CM, Hileman BM, Hutchinson AE, Chance EA, Huang GS. Perioperative hypoxemia is common with horizontal positioning during general anesthesia and is associated with major adverse outcomes: a retrospective study of consecutive patients. BMC Anesthesiol. 2014 Jun 9;14:43. doi: 10.1186/1471-2253-14-43. eCollection 2014. PMID 24940115
- [Background] Cotton BR, Smith G. The lower oesophageal sphincter and anaesthesia. Br J Anaesth. 1984 Jan;56(1):37-46. doi: 10.1093/bja/56.1.37. No abstract available. PMID 6140931
- [Background] Tiret L, Desmonts JM, Hatton F, Vourc'h G. Complications associated with anaesthesia--a prospective survey in France. Can Anaesth Soc J. 1986 May;33(3 Pt 1):336-44. doi: 10.1007/BF03010747. PMID 3719435
- [Background] Kozlow JH, Berenholtz SM, Garrett E, Dorman T, Pronovost PJ. Epidemiology and impact of aspiration pneumonia in patients undergoing surgery in Maryland, 1999-2000. Crit Care Med. 2003 Jul;31(7):1930-7. doi: 10.1097/01.CCM.0000069738.73602.5F. PMID 12847385
- [Background] Kluger MT, Short TG. Aspiration during anaesthesia: a review of 133 cases from the Australian Anaesthetic Incident Monitoring Study (AIMS). Anaesthesia. 1999 Jan;54(1):19-26. doi: 10.1046/j.1365-2044.1999.00642.x. PMID 10209365
- [Background] Ewig S, Torres A. Prevention and management of ventilator-associated pneumonia. Curr Opin Crit Care. 2002 Feb;8(1):58-69. doi: 10.1097/00075198-200202000-00010. PMID 12205408
- [Background] Torres A, Serra-Batlles J, Ros E, Piera C, Puig de la Bellacasa J, Cobos A, Lomena F, Rodriguez-Roisin R. Pulmonary aspiration of gastric contents in patients receiving mechanical ventilation: the effect of body position. Ann Intern Med. 1992 Apr 1;116(7):540-3. doi: 10.7326/0003-4819-116-7-540. PMID 1543307
- [Background] Reali-Forster C, Kolobow T, Giacomini M, Hayashi T, Horiba K, Ferrans VJ. New ultrathin-walled endotracheal tube with a novel laryngeal seal design. Long-term evaluation in sheep. Anesthesiology. 1996 Jan;84(1):162-72; discussion 27A. doi: 10.1097/00000542-199601000-00019. PMID 8572330
- [Background] Petring OU, Adelhoj B, Jensen BN, Pedersen NO, Lomholt N. Prevention of silent aspiration due to leaks around cuffs of endotracheal tubes. Anesth Analg. 1986 Jul;65(7):777-80. PMID 3717617
- [Background] Seegobin RD, van Hasselt GL. Aspiration beyond endotracheal cuffs. Can Anaesth Soc J. 1986 May;33(3 Pt 1):273-9. doi: 10.1007/BF03010737. PMID 3719428
- [Background] Smith G, Ng A. Gastric reflux and pulmonary aspiration in anaesthesia. Minerva Anestesiol. 2003 May;69(5):402-6. PMID 12768174
- [Background] Ferrer R, Artigas A. Clinical review: non-antibiotic strategies for preventing ventilator-associated pneumonia. Crit Care. 2002 Feb;6(1):45-51. doi: 10.1186/cc1452. Epub 2001 Jan 11. PMID 11940265
- [Background] Keenan SP, Heyland DK, Jacka MJ, Cook D, Dodek P. Ventilator-associated pneumonia. Prevention, diagnosis, and therapy. Crit Care Clin. 2002 Jan;18(1):107-25. doi: 10.1016/s0749-0704(03)00068-x. PMID 11910725
- [Background] Koeman M, van der Ven AJ, Ramsay G, Hoepelman IM, Bonten MJ. Ventilator-associated pneumonia: recent issues on pathogenesis, prevention and diagnosis. J Hosp Infect. 2001 Nov;49(3):155-62. doi: 10.1053/jhin.2001.1073. No abstract available. PMID 11716631
- [Background] Fernandez-Crehuet R, Diaz-Molina C, de Irala J, Martinez-Concha D, Salcedo-Leal I, Masa-Calles J. Nosocomial infection in an intensive-care unit: identification of risk factors. Infect Control Hosp Epidemiol. 1997 Dec;18(12):825-30. PMID 9442407
- [Background] Drakulovic MB, Torres A, Bauer TT, Nicolas JM, Nogue S, Ferrer M. Supine body position as a risk factor for nosocomial pneumonia in mechanically ventilated patients: a randomised trial. Lancet. 1999 Nov 27;354(9193):1851-8. doi: 10.1016/S0140-6736(98)12251-1. PMID 10584721
- [Background] Kollef MH. Ventilator-associated pneumonia. A multivariate analysis. JAMA. 1993 Oct 27;270(16):1965-70. PMID 8411554
- [Background] Institute for Healthcare Improvement: Prevent ventilator-associated pneumonia. Institute for Healthcare Improvement. 2012. http://www.ihi.org/knowledge/Pages/Changes/ImplementtheVentilatorBundle.aspx; Accessed 9 Dec 2013.
- [Background] Blitt CD, Gutman HL, Cohen DD, Weisman H, Dillon JB. "Silent" regurgitation and aspiration during general anesthesia. Anesth Analg. 1970 Sep-Oct;49(5):707-13. No abstract available. PMID 5534428
- [Background] McEwen DR. Intraoperative positioning of surgical patients. AORN J. 1996 Jun;63(6):1059-63, 1066-79; quiz 1080-6. doi: 10.1016/s0001-2092(06)63293-6. PMID 8771317
- [Background] Adedeji R, Oragui E, Khan W, Maruthainar N. The importance of correct patient positioning in theatres and implications of mal-positioning. J Perioper Pract. 2010 Apr;20(4):143-7. doi: 10.1177/175045891002000403. PMID 20446625
- [Background] Smith KA. Positioning principles. An anatomical review. AORN J. 1990 Dec;52(6):1196-202, 1204, 1206-8. doi: 10.1016/s0001-2092(07)69197-2. No abstract available. PMID 2278485
- [Background] Mulier JP, Dillemans B, Van Cauwenberge S. Impact of the patient's body position on the intraabdominal workspace during laparoscopic surgery. Surg Endosc. 2010 Jun;24(6):1398-402. doi: 10.1007/s00464-009-0785-8. Epub 2010 Jan 7. PMID 20054583
- [Background] Abdulla S. Pulmonary aspiration in perioperative medicine. Acta Anaesthesiol Belg. 2013;64(1):1-13. PMID 23767172
- [Background] Engelhardt T, Webster NR. Pulmonary aspiration of gastric contents in anaesthesia. Br J Anaesth. 1999 Sep;83(3):453-60. doi: 10.1093/bja/83.3.453. No abstract available. PMID 10655918
- [Background] Ng A, Smith G. Gastroesophageal reflux and aspiration of gastric contents in anesthetic practice. Anesth Analg. 2001 Aug;93(2):494-513. doi: 10.1097/00000539-200108000-00050. PMID 11473886
- [Background] Kalinowski CP, Kirsch JR. Strategies for prophylaxis and treatment for aspiration. Best Pract Res Clin Anaesthesiol. 2004 Dec;18(4):719-37. doi: 10.1016/j.bpa.2004.05.008. PMID 15460555
- [Derived] Michael Dunham C, Hileman BM, Hutchinson AE, Antonaccio T, Chance EA, Huang GS, Szmaj G, Calabro K, Bishop C, Schrickel TT. Evaluation of operating room reverse Trendelenburg positioning and its effect on postoperative hypoxemia, aspiration, and length of stay: a retrospective study of consecutive patients. Perioper Med (Lond). 2017 Aug 22;6:10. doi: 10.1186/s13741-017-0067-2. eCollection 2017. PMID 28852473